CLINICAL TRIAL: NCT01362881
Title: A Prospective Cohort Study of the Surgical Treatment of Early Onset Scoliosis Using a Remotely Expandable Device for Non-invasive Lengthening of a Growing Rod (Magec™) and Its Performance in Prevention of Progression of Scoliosis.
Brief Title: Study of the Surgical Treatment of Early Onset Scoliosis Using a Non-invasive Growing Rod
Status: Completed | Type: Observational
Sponsor: Ellipse Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SC-11-001
Record Dates: First submitted 2011-05-27; First posted 2011-05-30 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-06

CONDITIONS: Scoliosis
Keywords: Early; Onset; Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
It is current practice for children who have surgery for early onset scoliosis (EOS) to be treated with insertion of extendable implants known as growth rod systems. This allows the growth potential of the child to be maximised during the period of growth. However, the child must undergo an average of 6 further surgeries to lengthen the rods every 6 months. Sometimes this may continue for several years. This requires repeated general anaesthesia and places the patient at risk of complications as well as on-going costs to the hospital with each admission and theatre episode.

Magec is a magnetic growth rod from Ellipse technologies (distributed by SurgiC). The rod is inserted in exactly the same way as the conventional growth rod systems. The base implants i.e screws and hooks remain the preferred choice of the user. The only change is that a different rod is used.

There are several advantages to this device. Firstly, after the initial insertion, further lengthenings, unlike current systems, do not need to be carried out in theatre under a general anaesthetic. In contrast, they can be done in an outpatients setting with a non-invasive technique. The rods are lengthened using an external magnetic device. The lengthenings are done in a controlled manner using an age related growth guide. Thirdly, the change from a theatre based intervention to an outpatient procedure will have cost-savings. The investigators also believe that there will be psychosocial benefits to the child and family by the avoiding the stress associated with repeated surgery at such a young age.

In terms of risk assessment the device does not place the child at any more risk than would be expected from inserting any of the existing systems. In the event of failure of the rods the worst outcome is a revision to conventional rods.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 2 - 10 years (male/female) with EOS and growth potential
2. Patient who surgeon feels would benefit from the implantation of a growth rod
3. Patient must be of appropriate size and age for use of the device
4. Patient's guardian is willing and able to give informed consent for participation in the study
5. Patient (and guardian) is willing and able to return for all follow-up visits and study related procedures
6. The patient's guardian is willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study

Exclusion Criteria:

* The participant may not enter the study if ANY of the following apply:

  1. Conversion patients with prior construct problems
  2. Previous diagnosis of post-operative spinal infection or wound complication
  3. Conversion patients with more than 3 previous distractions, or more than 2 years since initial surgery
  4. Patients with prior failure of other devices
  5. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study
  6. Participants who have participated in another research study involving an investigational product in the past 12 weeks

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study population will be recruited from secondary care
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
To Assess the Safety and effectiveness of a Magnetic Growth Rod | 2 Years From Final Recruitment Date

CONTACTS AND LOCATIONS:
Overall Officials: Colin Nnadi, Principal Investigator — Consultant Surgeon
Locations (2):
- United Kingdom (2):
  - Leeds Teaching Hospitals, Leeds
  - Oxford University NHS Trust, Oxford

REFERENCES:
- See also: Oxford Spine Unit — http://www.ouh.nhs.uk/spinal/
- See also: Oxford University R&D — http://www.ouh.nhs.uk/researchers/